CLINICAL TRIAL: NCT07291895
Title: A Prospective Single-blinded Randomized Study of High Dose Radiotherapy for Palliation: Hi-D
Brief Title: High Dose Radiotherapy for Palliation (Hi-D)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hi-D
Record Dates: First submitted 2025-11-24; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Metastases; Palliative Radiotherapy
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Dose RT (Experimental): 27Gy in 3 fractions with boost
  Interventions: Radiation: Palliative Radiotherapy
- Standard Dose Palliative RT (Active Comparator): 24Gy in 3 fractions
  Interventions: Radiation: Palliative Radiotherapy

INTERVENTIONS:
Radiation: Palliative Radiotherapy — standard dose RT
  Arms: Standard Dose Palliative RT
Radiation: Palliative Radiotherapy — high-dose RT
  Arms: High-Dose RT

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility of single-blind randomization between two palliative regimens - standard 24 Gray in 3 fractions vs a high-dose (Hi-D) 27 Gray in 3 fractions with dose escalation within the tumor in participants with bulky metastatic cancer.

The main question

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all the following criteria to be eligible for participation in this study:
* Age 18 or older.
* Able to provide informed consent
* Patient has histologically confirmed solid tumour malignancy
* ECOG performance status 0 - 2
* Life Expectancy > 6 months
* 1-5 target lesions larger than 5cm
* A history and physical exam, including ECOG performance status, performed within 6 weeks prior to trial enrollment
* Not suitable for or declined curative-intent treatment
* Subject has had a CT neck, chest, abdomen and pelvis or PET-CT within 8 weeks prior to enrollment, and with 12 weeks of treatment
* MRI spine for patients receiving RT to vertebral or paraspinal metastases
* Patient is judged able to:

  * Maintain a stable position during therapy
  * Tolerate immobilization device(s) that may be required to deliver radiation safely

Exclusion Criteria:

* - Hematologic malignancy.
* Disease limited to intracranial sites
* Serious medical co-morbidities precluding radiotherapy
* Bone metastases with no soft tissue component
* Prior radiation to target lesion that precludes delivery of repeat radiation. All such cases should be discussed with the local and study PIs.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of accrual | From open to accrual to close to accrual (24 months)
  ≥20 participants enrolled within 24 months from first patient accrued
Feasibility of blinding | From enrollment to RT completion.
  Trial Assignment Questionnaire administered post-treatment.

SECONDARY OUTCOMES:
Compare changes in local control | From enrollment to end of study, accessed at 6 weeks, and month 3,12,18,24
  Kaplan-Meier curves; stratified log-rank test
Compare changes in OS | From enrollment to end of study at 24 months or death
  Time from randomization to death from any cause. Kaplan-Meier; stratified log-rank.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Liu, MD, FRCPC, Principal Investigator — BC Cancer - Vancouver
Locations (1):
- BC Cancer - Vancouver, Vancouver, British Columbia, Canada